CLINICAL TRIAL: NCT02166229
Title: Divalproex Sodium in the Treatment of the Cutaneous Manifestations of Scleroderma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No subjects were enrolled.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1404013775
Record Dates: First submitted 2014-06-10; First posted 2014-06-18 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Scleroderma; Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Divalproex sodium (Experimental): Divalproex sodium will be initiated at 125 mg twice daily and increased monthly to a maximum dose of 500 mg twice daily.
  Interventions: Drug: Divalproex sodium

INTERVENTIONS:
Drug: Divalproex sodium

SUMMARY:
To investigate the ability of divalproex sodium, a histone deacetylase inhibitor, to improve the digital manifestations of scleroderma including digital edema, calcinosis cutis, digital ulcers, and joint contractures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of scleroderma as defined by the American College of Rheumatology (ACR)
* Presence of at least one digital manifestation occurring within the past 6 months, i.e. digital swelling/edema, digital ulcer, calcinosis cutis, restricted digital range of motion.
* Females of childbearing potential must take an oral contraceptive pill or use an equivalent birth control method during the study.

Exclusion Criteria:

* Age <18 years old
* Ongoing use of high dose steroids (>10 mg/day) or unstable steroid dose in past 4 weeks.
* An investigational drug or disease-modifying agent has been started within the past 6 months, including but not limited to systemic corticosteroids, methotrexate, cyclosporine, azathioprine, cyclophosphamide, bosentan, mycophenolate mofetil, thalidomide, colchicine.
* Patient taking a medication with a significant drug-drug interaction with divalproex sodium, e.g. clomipramine and lamotrigine.
* Patient has another connective tissue disease or other condition that could affect rest pain and hand function, e.g. systemic lupus erythematosus, rheumatoid arthritis, or osteoarthritis.
* Patient has uncontrolled diabetes, chronic kidney disease, chronic hepatitis.
* Any of the following laboratory abnormalities at baseline: anemia (Hb < 8.5 gm/dL), thrombocytopenia with platelets <100,000, INR > 1.3 or known bleeding disorder, estimated GFR < 60 mL/min/1.73m2 or serum creatinine > 2.0 mg/dL, hyperbilirubinemia or elevation of AST or ALT
* Pregnancy or breast-feeding.
* History of severe depression (i.e. depression requiring medical treatment by a psychiatrist), suicidal ideation, epilepsy, bipolar disorder, or schizophrenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of new digital ulcers | 12 months

SECONDARY OUTCOMES:
Change in modified Rodnan skin score | 12 months
Change in digital goniometry measurements | 12 months
  Goniometry measures range of motion of joints and, in this study, will include measurements of the metacarpophalangeal, proximal interphalangeal, distal interphalangeal and wrist joints.
Change in hydraulic pinch and hand-grip strength measurements | 12 months
Change in digital circumference | 12 months
Change in maximum oral aperture | 12 months
Change in estimated affected total body surface area | 12 months
Scleroderma Health Assessment Questionnaire (SHAQ) | 12 months
Number of new lesions of calcinosis cutis | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Brett King, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States